CLINICAL TRIAL: NCT03421704
Title: A Prospective Multicenter Registry of Patients With Sleep Disordered Breathing Treated With DreamStation BiPAP autoSV.
Acronym: autoSVREGDE
Status: Completed | Type: Observational
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Other Study IDs: SRC-SLE-ASVREGDE-2017-10032
Record Dates: First submitted 2018-01-10; First posted 2018-02-05 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Central Sleep Apnea; Mixed Sleep Apnea; Cheyne-Stokes Respiration; Complex Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Central; Sleep Apnea Syndromes; Cheyne-Stokes Respiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: DreamStation BiPAP autoSV — Philips Respironics DreamStation BiPAP autoSV (PR DS-autoSV) is designed to deliver pressure support for patient ventilatory assistance

SUMMARY:
This multi-center observational study will prospectively collect data from patients who have an indication for servo ventilation therapy. This registry is intended to characterize the patient populations that may benefit from DreamStation BiPAP autoSV therapy (PR DS-autoSV, Philips Respironics, Monroeville, PA) in real life settings. In addition, this registry will assess adherence to the PR DS-autoSV therapy, the therapeutic benefits, collect morbidity and mortality data of servo ventilation in patients with central sleep apnea (CSA) and complex sleep-disordered breathing (SDB).

ELIGIBILITY:
Inclusion Criteria:

* Indication and prescription of PR DS-autoSV
* Polysomnographic (PSG) or Polygraphic (PG) documentation of sleep-disordered breathing requiring servo ventilation

Exclusion Criteria:

* Patients with HFrEF - heart failure and low ejection fraction (EF ≤ 45%) and predominant CSA (> 50 % of events)
* Patients not able to receive positive airway pressure support through a mask due to surgical procedure or anatomical condition
* Chronic conditions with life expectancy < 1 year
* Significant chronic obstructive pulmonary disease (COPD) with an FEV1/VC < 70% (GOLD III)
* Respiratory insufficiency requiring long-term oxygen therapy
* Daytime hypercapnia at rest (pCO2 > 45 mmHg)
* Cardiac surgery, PCI, myocardial infarction, unstable angina, within 12 weeks prior to enrolment
* Cardiac resynchronization or pacemaker implantation within the last 6 months
* Untreated or therapy refractory Restless legs-Syndrome (RLS)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry will include adult participants with indication and prescription of PR DS-autoSV
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Short term Device usage and therapy adherence | 6 months
  Device usage (hours/ night). Patients will be classified into various adherence subgroups based on the average daily device use at each study interval. The percentage of participants in each of the adherence subgroups will be presented.

SECONDARY OUTCOMES:
Long term Device usage and therapy adherence | 12 months
  EDevice usage (hours/ night). Patients will be classified into various adherence subgroups based on the average daily device use at each study interval. The percentage of participants in each of the adherence subgroups will be presented.
Change in Health-related quality of life | 6, 12 and 24 months
  European Quality of Life-5 Dimensions questionnaire EQ 5D- 5L) is a standardized instrument for measuring generic health related quality of life. This tools scores range from 1 to 5, with higher scores indicating more problems across five dimensions (5D) which comprise mobility, self-care, usual activities, pain/discomfort, and anxiety/depression
Change in Subjective sleep quality | 6, 12 and 24 months
  Pittsburgh Sleep Quality Index (PSQI)
Change in Daytime sleepiness. | 6, 12 and 24 months
  Epworth Sleepiness Scale (ESS). This test consists of eight questions of daily life activities with a number from 0 (not at all likely to fall asleep) to 3 (very likely to fall asleep) which yields a score of 0 to 24, and subjectively quantify sleepiness.25 An ESS score ranging from 0 to 10 is interpreted as normal, scores of 11 to 24 is considered to be abnormal and indicative of increasing levels of excessive daytime sleepiness.
Change on PSG/PG Parameters from baseline | 6 months
  Disordered breathing events
Change on PSG/PG Parameters from baseline | 6 months
  Quality of Sleep
Mortality | 6, 12 and 24 months
  Frequency of death in patients who showed adherence to therapy as compared to those with non-adherence
Causes of death | 6, 12 and 24 months
  causes of death , if available, will be compared in patients who showed adherence to therapy as compared to those with non-adherence
Number of healthcare utilization | 6, 12 and 24 months
  Number of hospitalizations during the minimum of one year follow-up, time to first hospitalization, composite number of unscheduled visits to emergency rooms and/or physician's office) in patients who showed adherence to therapy as compared to those with non-adherence (if data is available)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Arzt, MD, Principal Investigator — University Hospital Regensburg
Locations (9):
- Germany (9):
  - Universitätsklinikum der Ruhr-Universität Bochum, Bad Oeynhausen
  - Charité, Berlin
  - Klinik Donaustauf, Donaustauf
  - Helios Klinik Hagen Ambrok, Hagen
  - Muenster University Hospital, Münster
  - University Hospital Regensburg, Regensburg
  - Fachkrankenhaus Kloster, Schmallenberg
  - Helios Kliniken Schwerin, Schwerin
  - Wissenschaftliches Institut Bethanien für Pneumologie e.V, Solingen

IPD SHARING:
Plan to Share IPD: No